CLINICAL TRIAL: NCT04085731
Title: Driver-guided Ablation in the Treatment of Persistent Atrial Fibrillation
Brief Title: Driver-guided Ablation of Persistent Atrial Fibrillatiom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, Director, IRCCS Policlinico S. Donato
Other Study IDs: Persistent AF Ablation
Record Dates: First submitted 2019-09-07; First posted 2019-09-11 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheter ablation — Driver-guided catheter ablation of persistent atrial fibrillation

SUMMARY:
This is a prospective, single-center, study. A targeted number of 181patients with persistent AF will be included according to pre-defined criteria. The ablation procedure consists on the identification of the arrhythmic substrate using a novel integrated mapping technique. We hypothesize that such approach may potentially lead to a mechanisms-targeted ablation strategy of persistent AF.

DETAILED DESCRIPTION:
This is a prospective, single-center, study enrolling a total of 181patients with persistent AF according to well defined inclusion and exclusion criteria. The ablation procedure consists on the identification of the arrhythmic substrate using a novel integrated 3D mapping technique followed by standard CPVA at the end of the procedure. We will ablate substrates showing fast and regular electrical activities, starting from areas with the fastest mean cycle length and/or areas that have consistent rotational or focal propagation pattern and/or areas that comprise the slow conduction zone of possible arrhythmia circuits. After substrate ablation and AF termination, arrhythmia inducibility will be assessed and, if not inducible, the procedure will be completed by standard CPVA. If AF is still inducible, a new 3D map will be performed to identify further targets to be eliminated. Electrical cardioversion may be done at the end of the procedure. We hypothesized that such approach may potentially lead to a mechanisms-targeted ablation strategy leading to elimination of arrhythmic sources in individual patients, thus improving their clinical outcome. We will also characterize, identify and target the real pathophysiological substrates. After ablation, AF recurrence will be assessed by implantable loop recorder or thans-telephonic ECG recording from the end of the 3 months blanking period to 12 months following the procedure.The duration of this study is expected to be 24 months, from the first patient enrollment to the last patient follow-up.

ELIGIBILITY:
Inclusion Criteria: Age (18-85 years), persistent AF according to ESC/EHRA guidelines, first or second ablation procedure, ability to provide informed written consent.

-

Exclusion Criteria: Secondary AF, Hyperthyroidism, LVEF<30%, NYHA functional class IV, uncorrected valvular heart diseases, contraindication to anticoagulation, left atrial thrombus, recent (<6 months) myocardial infarction, thoracic surgery for congenital, valvular diseases, History of cerebrovascular events, pregnancy, cancer or other significant comorbidities.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 181 subjects suffering from persistent Atrial Fibrillation will be enrolled. Subject screening and enrollment will be carried out for approximately 12 months. A subject, who mets all of the inclusion criteria, and none of the exclusion criteria, is eligible to participate in this study. All patients will be accounted for and documented, assigning an identification code linked to their names, alternative identification, or contact information.This log will be kept up to date throughout the clinical study by the principal investigator. To ensure subject privacy and confidentiality of data this log must be maintained throughout the clinical study at the clinical site.
Sampling Method: Probability Sample
Enrollment: 181 (Estimated)
Dates: Start 2019-09-21 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from any AF or atrial tachycardia assessed from the end of the months blanking period to 12 months after ablation. | 12 months after ablation
  AF recurrences will be documented by implantable loop recorder or trns-telephonic ECG recording

SECONDARY OUTCOMES:
Identification of electrophysiological substrate | during the procedure
  Areas with fast but regular activities or with consistent wave front propagation pattern, or with low P-P voltage, or complex fractionated electrograms
inducibility of AF after the procedure | during the procedure
  programmed atrial stimulation before and after isoproterenol
AF burden | 12 months after ablation
  Assessment of AF burden by trans-telephonic ECG recording or implantable loop recorder

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — IRCCS San Donato University Hospital Policlinico San Donato, Milan, Italy
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided